CLINICAL TRIAL: NCT00003775
Title: A Phase II Open Label Study of SU101 for Patients With Anaplastic Astrocytoma in First Relapse
Brief Title: Leflunomide in Treating Patients With Anaplastic Astrocytoma in First Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: SUGEN-SU101.021; CDR0000066904; MSKCC-98111; NCI-G99-1506
Record Dates: First submitted 1999-11-01; First posted 2004-09-14 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult anaplastic astrocytoma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Astrocytoma; Glioma | interventions — Leflunomide

INTERVENTIONS:
Drug: leflunomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of leflunomide in treating patients who have anaplastic astrocytoma in first relapse.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the median time to progression, median survival, and objective response of patients with anaplastic astrocytoma or anaplastic oligoastrocytoma in first relapse treated with intravenous leflunomide (SU101). II. Assess the safety of SU101 in these patients. III. Describe the health-related quality of life of patients treated with intravenous SU101.

OUTLINE: This is an open label, multicenter study. Patients receive leflunomide (SU101) IV over 6 hours on days 1-4. Patients then receive SU101 IV over 6 hours weekly for 6 weeks (beginning between days 8-12). Patients exhibiting complete response, partial response, or stable disease may continue on treatment for up to a year or until disease progression or unacceptable toxicity occurs. Patients continuing therapy receive SU101 IV over 6 hours every week for 7 weeks, followed by 1 week of rest. Quality of life is assessed every 8 weeks and at the end of the study. Patients are followed every 8 weeks or until tumor progression.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed anaplastic astrocytoma or anaplastic oligoastrocytoma in first relapse Recurrence or progression at least 6 months from initial diagnosis Must have received maximally feasible surgical resection and fractionated external beam radiotherapy Must have received no more than 1 prior systemic cytotoxic chemotherapy regimen for initial disease Bidimensionally measurable disease by MRI scan (stable dose of corticosteroids for at least 7 days prior to scan)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 75,000/mm3 Hemoglobin at least 9 g/dL Hepatic: AST no greater than 3 times upper limit of normal (ULN) Bilirubin less than 1.5 times ULN Renal: Creatinine no greater than 2 mg/dL OR Creatinine clearance at least 40 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after the study No known allergy to etoposide No other acute or chronic medical illness or psychiatric disorder

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior epoetin alfa, filgrastim (G-CSF), or sargramostim (GM-CSF) and recovered No concurrent immunotherapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (2 weeks since vincristine; 6 weeks since nitrosoureas or mitomycin) and recovered No prior leflunomide (SU101) therapy No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy (except medroxyprogesterone acetate for appetite stimulation) Radiotherapy: See Disease Characteristics No more than 1 prior course of radiotherapy At least 8 weeks since prior radiotherapy and recovered No prior interstitial radiotherapy or implanted carmustine wafers Prior radiosensitizer(s) concurrent with radiotherapy or used as neoadjuvant therapy allowed No concurrent radiotherapy Surgery: See Disease Characteristics No more than 2 prior surgical resections At least 1 week since prior surgery or biopsy for anaplastic astrocytoma No concurrent surgery (including resection, stereotactic surgery, or interstitial implants) Other: At least 4 weeks since prior investigational agents No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1998-12; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison L. Hannah, MBBS, Study Chair — SUGEN
Locations (26):
- United States (22):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer Center of Albany Medical Center, Albany, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Neurological Institute, New York, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario